CLINICAL TRIAL: NCT04052750
Title: Daily Short Message Service Reminders Increase Treatment Compliance and Efficacy in Outpatients With Functional Gastrointestinal Disorders: a Randomized Controlled Trial
Brief Title: SMS Reminders and Treatment Compliance and Efficacy in Patients With FGIDs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shengliang Chen, professor,chief physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RJYYXHNK-004
Record Dates: First submitted 2019-08-03; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Functional Gastrointestinal Disorders; Patient Compliance
Keywords: Functional Gastrointestinal Disorders, Adherence
MeSH Terms: conditions — Gastrointestinal Diseases; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (No Intervention): Patients in this group only received medications without daily text message reminder
- The intervention group (Experimental): Patients in this group received a daily short message service (SMS) reminder when medications were prescribed
  Interventions: Behavioral: SMS follow-up

INTERVENTIONS:
Behavioral: SMS follow-up — In addition to conventional treatment, the experimental group received SMS reminding every day until the end of the treatment.
  Arms: The intervention group

SUMMARY:
The effect of SMS follow-up on drug compliance and efficacy in patients with FGIDs has not been reported in the literature. We, therefore, conducted a prospective randomized controlled trial to investigate whether SMS follow-up could improve treatment adherence in patients with FGIDs, which in turn would help symptom relief and improve treatment outcomes.

DETAILED DESCRIPTION:
The irritable bowel syndrome (IBS) and other functional gastrointestinal disorders (FGIDs) are common and pose significant burdens to patients. Although regular medications have substantial benefits for disease remission, many patients do not follow the recommendations of standard medication regimens given by physicians at the time of the visit, so how to improve patient compliance becomes even more important. Many factors can affect drug compliance. Forgetting seems to be one of the important reasons for poor compliance. In order to solve this problem, many studies such as drug charts/calendars, mini kits, etc. have been conducted in previous studies. At present, with the popularization of mobile phones, SMS-based interventions are gradually being applied to various medical environments. Compared with the phone, SMS consumes less time and can be easily integrated into the patient's daily life. Therefore, short messages may be more suitable for follow-up of patients outside hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed FGIDs according to Rome-IV
* Aged 18-70 years
* With no obvious organic abnormalities

Exclusion Criteria:

* With organic gastrointestinal diseases
* With psychiatric diseases or are taking psychotropic agents
* With severe cardiopulmonary or other organ diseases
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Treatment compliance in outpatients with FGIDs | week2
  Compliance is assessed by the medication possession ratio (MPR). The MPR is often defined as the sum of the days' supply of medication divided by the number of days between the first fill and the last refill plus the days' supply of the last refill. This calculation usually results in a ratio less than 1.0 if there are lapses in prescription refilling.

SECONDARY OUTCOMES:
Improvement of abdominal pain in outpatients with FGIDs | week2
  Improvement of abdominal pain symptom was assessed by comparison of symptom score after treatment to that before treatment. The pain symptome was assessed by Visual Analog Score for pain with the following creteria: 0, no pain; 1, mild; 2, related; 3, severe; 4, very severe. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- RenJiH, Shanghai, China

REFERENCES:
- [Derived] Wang B, Luo QQ, Li Q, Cheng L, Chen SL. Daily Short Message Service Reminders Increase Treatment Compliance and Efficacy in Outpatients with Functional Dyspepsia: a Prospective Randomized Controlled Trial. J Gen Intern Med. 2020 Oct;35(10):2925-2931. doi: 10.1007/s11606-020-06088-3. Epub 2020 Aug 10. PMID 32779141